CLINICAL TRIAL: NCT01832168
Title: A Prospective Randomized Clinical Trial Using Amniotic Membrane in Robotic Assisted Laparoscopic Prostatectomy (RALP)- Effect on Nerve Protection.
Brief Title: Randomized Clinical Trial Using Amniotic Membrane in Robotic Assisted Laparoscopic Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFRALP001
Record Dates: First submitted 2013-04-11; First posted 2013-04-15 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Pudendal Nerve

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Other): Robotic Assisted Laparoscopic Prostatectomy with application of absorbable hemostat.
  Interventions: Procedure: Robotic Assisted Laparoscopic Prostatectomy; Other: Application of Absorbable Hemostat
- AmnioFix (Experimental): Robotic Assisted Laparoscopic Prostatectomy with application of dehydrated human amniotic membrane.
  Interventions: Procedure: Robotic Assisted Laparoscopic Prostatectomy; Other: Application of dehydrated human amniotic membrane

INTERVENTIONS:
Procedure: Robotic Assisted Laparoscopic Prostatectomy — Robotic Assisted Laparoscopic Prostatectomy with nerve-sparing technique
Other: Application of Absorbable Hemostat — Application of Surgicel® SNoW Absorbable Hemostat by Johnson and Johnson on the neurovascular bundle after removal of the cancerous prostate.
  Other Names: Surgicel® SNoW
  Arms: Control
Other: Application of dehydrated human amniotic membrane — Application of dehydrated human amniotic membrane (DHAM) on the neurovascular bundle after removal of the cancerous prostate.
  Other Names: AmnioFix
  Arms: AmnioFix

SUMMARY:
The purpose of this study is to determine whether the AmnioFix dehydrated human amniotic membrane is effective in protecting nerves in men receiving robotic assisted laparoscopic prostatectomies.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 45-70
2. Clinically localized prostate cancer with Gleason score 6 or 7
3. SHIM Score greater than or equal to 16 in the absence of medication
4. Feasibility to perform unilateral or bilateral nerve sparing RALP

Exclusion Criteria:

1. Clinically locally advanced cancer and/or with Gleason score 8 or 9.
2. Difficulty performing nerve sparing RALP.
3. Prior surgery at the site.
4. Site exhibits clinical signs and symptoms of infection.
5. SHIM score at screening <16.
6. Current use of anticoagulant medication including Coumadin, Plavix, etc.
7. Has had "salvage prostatectomy" - patients who failed prior therapies including external radiation therapy, cryotherapy, etc.
8. Has prior radiation therapy treatment at the site.
9. Prior hormonal therapy such as Lupron or oral anti-androgens.
10. Non-mobile, i.e. not ambulatory or bed ridden.
11. The presence of comorbidities that can be confused with or can exacerbate the condition including:

    1. diabetes
    2. advanced atherosclerotic vascular disease
12. Patients with a history of more than two weeks treatment with immuno-suppressants (including systemic corticosteroids), cytotoxic chemotherapy within one month prior to initial screening, or who receive such medications during the screening period, or who are anticipated to require such medications during the course of the study.
13. Patients on any investigational drug(s) or therapeutic device(s) within 30 days preceding screening.
14. Unable to comply with penile rehabilitation.
15. Known history of having Acquired Immunodeficiency Syndrome (AIDS) or HIV.
16. Patients who are unable to understand the aims and objectives of the trial.
17. Presence of any condition(s) which seriously compromises the subject's ability to complete this study, or has a known history of poor adherence with medical treatment.
18. Currently taking medications which could affect graft incorporation (supervising physician's discretion).
19. Allergic to gentamicin and/or streptomycin.
20. Damage to neurovascular bundles during surgery.

Ages: 45 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The proportion of patients achieving return to baseline Sexual Health Inventory for Men (SHIM) score in the AmnioFix group versus the Control group. | 4 weeks

SECONDARY OUTCOMES:
Time to return of erectile function. | Up to 6 months
Pain scores. | 10 days, 4 weeks, 3 months, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Razdan, MD, Principal Investigator — Jackson South Urology Center of Excellence
Locations (1):
- Jackson South Urology Center of Excellence, Miami, Florida, United States